CLINICAL TRIAL: NCT04274556
Title: Do Biochemical Parameters and Intradialytic Symptoms Affect Post-dialysis Recovery Time?: A Cross-sectional Study
Brief Title: Recovery Time and Affecting Factors in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Assistant Professor, Istanbul Demiroglu Bilim University
Other Study IDs: 03
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Dialysis; Complications; Life Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Post-dialysis recovery group — Before the hemodialysis session, the patients were asked by the investigators how long it took them to recover from a dialysis session, taking the last treatment month into account.

SUMMARY:
Patients undergoing hemodialysis (HD) can experience symptoms such as lassitude, pain, muscle cramps, nausea, vomiting, constipation, diarrhea, rash, skin dryness, sleep disorders, and emotional and sexual problems after the treatment. Many chronic HD patients do not feel well after the treatment sessions and need some time to recover. This recovery time is defined as the time required to recover from the feelings of lassitude and fatigue.

DETAILED DESCRIPTION:
The recovery time not only decreases the quality of life but also increases the risk of mortality and morbidity. As a prolonged recovery time affects both the patients and the healthcare professionals and caregivers, there has been increased interest on determining the modifiable treatment-related factors in the international literature. The patients are limited in their daily living activities at home and at work during this period and a significant amount of time is therefore required to go back to normal life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Being on HD for 4 hours a day on 3 days per week for at least 6 months
* No communication problem
* Volunteering to participate to the study

Exclusion Criteria:

* Younger than 18 years
* Shorter being on HD for 4 hours a day on 3 days per week for at least 6 months
* Have communication problem
* Not volunteering to participate to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being on HD for 4 hours a day on 3 days per week for at least 6 months and 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Demiroglu Bİlim University, Istanbul, Sisli
  - Demiroglu Bilim University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bossola M, Di Stasio E, Antocicco M, Silvestri P, Tazza L. Variables associated with time of recovery after hemodialysis. J Nephrol. 2013 Jul-Aug;26(4):787-92. doi: 10.5301/jn.5000198. Epub 2012 Aug 31. PMID 22941875
- [Background] Bossola M, Marzetti E, Di Stasio E, Monteburini T, Cenerelli S, Mazzoli K, Parodi E, Sirolli V, Santarelli S, Ippoliti F, Nebiolo PE, Bonomini M, Melatti R, Vulpio C. Prevalence and associated variables of post-dialysis fatigue: Results of a prospective multicentre study. Nephrology (Carlton). 2018 Jun;23(6):552-558. doi: 10.1111/nep.13059. PMID 28419668
- [Background] Davenport A, Guirguis A, Almond M, Day C, Chilcot J, Wellsted D, Farrington K. Comparison of characteristics of centers practicing incremental vs. conventional approaches to hemodialysis delivery - postdialysis recovery time and patient survival. Hemodial Int. 2019 Jul;23(3):288-296. doi: 10.1111/hdi.12743. Epub 2019 Mar 12. PMID 30860667
- [Derived] Ozen N, Cepken T, Tosun B. Do biochemical parameters and intradialytic symptoms affect post-dialysis recovery time? A prospective, descriptive study. Ther Apher Dial. 2021 Dec;25(6):899-907. doi: 10.1111/1744-9987.13624. Epub 2021 Feb 8. PMID 33497021

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-dialysis Recovery Group
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Post-dialysis Recovery Group
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-dialysis Recovery Time
Description: Before the hemodialysis session, the patients were asked by the investigators how long it took them to recover from a dialysis session, taking the last treatment month into account.
Time Frame: Up to 7 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Post-dialysis Recovery Group
Number analyzed (Participants) | 86
minutes | 278.02 (209.94)

2. Primary Outcome: Number of Participants With Intradialytic Hypotension
Description: It is defined in the European Best Practice Guideline (EBPG) as a decrease of 20 mmHg or more in the systolic blood pressure or 10 mmHg or more in the mean arterial blood pressure together with symptoms requiring nursing intervention.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Post-dialysis Recovery Group
Number analyzed (Participants) | 86
Participants
  Existing of intradialytic symptoms | 42
  Absent of intradialytic symptoms | 44

3. Primary Outcome: Rate of Dialysis Symptoms
Description: It was identified with Dialysis Symptom Index (DSI). DSI consists of 30 items. We queried the subjects regarding symptoms in the last 7 days. The effect was evaluated with a Likert type scale from 0 to 4, representing "not at all" to "significantly". The total score of the DSI ranges from 0 to 150. A score of zero reflects no symptoms while increasing total scores reflect increasing effects of the symptoms.
Time Frame: Up to 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-dialysis Recovery Group
Number analyzed (Participants) | 86
score on a scale | 19.10 (14.29)

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Description: Side effects/other adverse events were not monitored
Arm/Group | Post-dialysis Recovery Group
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT04274556/Prot_SAP_000.pdf